CLINICAL TRIAL: NCT06989138
Title: The Effect of Orthosis and Exercise Training on Pain, Physical Function and Quality of Life in Patients With Spondylolisthesis
Brief Title: Effects of Orthosis & Exercise on Spondylolisthesis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: Baltalimani Bone Diseases Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Fatma Dilge ASIK BOZDEMIR, Lecturer - PhD(c), Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-2220
Record Dates: First submitted 2025-05-05; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Spondylolisthesis; Orthosis; Exercise Training
Keywords: Spondylolisthesis; Orthosis; Exercise; Stabilization; Physical function; Kinesiophobia
MeSH Terms: conditions — Spondylolisthesis; Motor Activity; Kinesiophobia | interventions — Orthotic Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stabilization Exercise Group (Experimental): Participants diagnosed with spondylolisthesis after randomization and assigned to the stabilization exercise group will be treated after being evaluated by the research therapist. In this context, the physiotherapist will structure a program consisting of a combination of recommended soft orthosis, pain control, stabilization exercises, posture training and home exercises. Soft orthosis will be applied for 10-12 hours a day for 4-6 weeks; 20 minutes of TENS and 20 minutes of Hotpack for pain control; and stabilization exercises with Stabilizer Pressure Biofeedback device. The planned stabilization exercise program will be 30-35 minutes; 15 minutes of posture training will be applied. These applications will be performed in the clinical environment 2 days a week for 10 weeks with a physiotherapist. Participants will be asked to practice the home exercise program taught in the training session 6 days a week for 12 weeks, excluding clinical applications.
  Interventions: Other: Stabilitation Exercise; Other: Orthosis
- Conventional Exercise Group (Experimental): After randomization, participants assigned to the conventional exercise group and diagnosed with spondylolisthesis will be evaluated and treated by the research therapist. In this context, the physiotherapist will structure a program consisting of a combination of the recommended soft orthosis, physiotherapy (pain control and exercise) and home exercises. The soft orthosis will be applied 10-12 hours a day for 4-6 weeks; 20 minutes of TENS and 20 minutes of Hotpack for pain control; 30-35 minutes of conventional exercise program will be applied. These applications will be performed in the clinical environment 2 days a week for 10 weeks in the presence of a physiotherapist. Participants will be asked to perform the home exercise program taught in the training session 6 days a week for 12 weeks, excluding clinical applications.
  Interventions: Other: Conventional Exercise; Other: Orthosis
- Control Group (No Intervention): Individuals who have been diagnosed with spondylolisthesis and have not undergone the recommended treatment will be included in the control group for the study.

INTERVENTIONS:
Other: Stabilitation Exercise — Patients will be included with the guidance of a physician specialized in the relevant field. After randomization, the patients included in the groups will be given 1 session of training before the start of treatment. In this training, soft orthosis use and home exercise programs will be explained to the patients in the intervention group. Soft orthoses; It will be explained that they should use for 10-12hours during the day for 4-6weeks, take them off during rest, sleep and exercise, and use them during active hours. Home exercise program; as in the classical approach, stretching and strengthening exercises will first be explained to the patient practically by the physiotherapist and then the patient will be asked to practice. Participants will be accompanied by a physiotherapist in the clinical environment 2 days a week for 10 weeks according to the groups they are divided into. Patients will be asked to practice the home exercise program taught in the training session 6 days a week.
  Arms: Stabilization Exercise Group
Other: Conventional Exercise — Patients will be included with the guidance of a physician specialized in the relevant field. After randomization, the patients included in the groups will be given 1 session of training before the start of treatment. In this training, soft orthosis use and home exercise programs will be explained to the patients in the intervention group. Soft orthoses; It will be explained that they should use for 10-12hours during the day for 4-6weeks, take them off during rest, sleep and exercise, and use them during active hours. Home exercise program; as in the classical approach, stretching and strengthening exercises will first be explained to the patient practically by the physiotherapist and then the patient will be asked to practice. Participants will be accompanied by a physiotherapist in the clinical environment 2 days a week for 10 weeks according to the groups they are divided into. Patients will be asked to practice the home exercise program taught in the training session 6 days a week.
  Arms: Conventional Exercise Group
Other: Orthosis — Patients will be included with the guidance of a physician specialized in the relevant field. After randomization, the patients included in the groups will be given 1 session of training before the start of treatment. In this training, soft orthosis use and home exercise programs will be explained to the patients in the intervention group. Soft orthoses; It will be explained that they should use for 10-12hours during the day for 4-6weeks, take them off during rest, sleep and exercise, and use them during active hours.
  Arms: Conventional Exercise Group; Stabilization Exercise Group

SUMMARY:
In the treatment of spondylolisthesis, conservative methods are initially preferred unless severe neurological symptoms are present; surgical treatment is only performed in refractory cases lasting at least 3-6 months. Conservative treatment consists of orthotic use, activity restriction, pain control, physiotherapy and exercise. Orthotics may promote healing by restricting movement; however, there are not enough studies on this subject. Exercise is the intervention with the highest level of evidence in chronic low back pain. The efficacy of stabilisation exercises in providing positive and long-lasting effects on pain and functional disability in patients with spondylolisthesis has been demonstrated. However, studies evaluating the effect of exercise on spinal stability and radiological findings are limited. Therefore, this study aims to compare the effects of stabilization and conventional exercises with orthosis on radiographic findings, pain, physical function and quality of life.

DETAILED DESCRIPTION:
Treatment is initially conservative (in the absence of severe neurologic symptoms) and surgical treatment is only indicated for those who have been refractory to non-surgical options for at least 3 to 6 months. Conservative treatment usually consists of orthotics, activity restriction, pain control, physiotherapy program and exercise. It has been reported in the literature that the use of orthotics helps to restrict activities by acting as a physical barrier against provocative movements and allows sufficient immobilization to promote healing. However, there are not enough studies on this subject in the literature. Exercise is the intervention with the highest level of evidence for improving CLBP and is superior to all other interventions in terms of improving pain and function.

In the literature, it has been reported that stabilization exercises, one of the current types of exercises recommended for patients with spondylolisthesis, can reduce pain and functional disability in patients and that this effect can be maintained over a 30-month follow-up period. There are a limited number of studies investigating whether exercise therapy can objectively contribute to the improvement of structural stability and intervertebral motion in the spine, especially in patients with grade-I slippage preferably managed with non-invasive treatments, and the effect of exercise therapy on radiological findings in patients affected by spondylolisthesis. In the light of this information, it was planned to compare the effects of stabilization and conventional exercises combined with orthosis use on radiographic findings, pain level, physical function and quality of life in patients with spondylolisthesis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65
* Individuals without indication for surgery
* Individuals diagnosed with grade 1-2 spondylolysis
* Individuals without neurological deficits
* Individuals diagnosed with radicular pain or non-specific chronic low back pain for more than 3 months

Exclusion Criteria:

* Surgery recommended after diagnosis
* History of lumbar surgery
* Presence of rheumatic inflammatory diseases or diabetic polyneuropathy
* Individuals with symptoms of cauda equina or ischemic heart disease
* Presence of back pain with non-mechanical causes or non-radicular neuropathic pain
* Having received this type of exercise therapy before

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life Scale Short Form | Week 0, week 10, week 12
  The scale, consists of 4 sections (physical health, psychological health, social relations and environment) and a total of 27 questions. The individual is asked to score the questions between 1-5, taking into account the last 15 days. Higher scores in the total score and subscales indicate better quality of life.
Berg Balance Scale | Week 0, week 10, week 12
  This scale is a 14-question test assessing postural control and fall risk. Each question is scored between 0-4 and the maximum score is 56. 0-20 points are defined as impaired balance / high fall risk, 21-40 points as acceptable balance / moderate fall risk, 41-56 points as good balance / low fall risk.
Joint Position Sensation | Week 0, week 10, week 12
  It will be assessed by joint position sense, which measures the patients' ability to actively reposition the lower back to their neutral position. The patient will be seated with feet on the floor, hands on the thighs, hip-knee flexed 90 degrees with the back on a hard surface and the patient will be instructed to assume a neutral lumbar spine position. The stabilizer pressure biofeedback device will be placed between the neutral spine and the hard surface and inflated to 70 mmHg. The participant will be asked to perform maximal anterior and posterior pelvic tilts 2 times in succession, waiting 5 seconds at each end point, and then return to the neutral position. The pressure difference between the initial and final measurement will be recorded.
McGill Pain Questionnaire Short Form | Week 0, week 10, week 12
  In the questionnaire, pain level is defined with 15 words consisting of 11 sensory and 4 affective words (0-3 points). The pain felt at the time of the questionnaire is measured with the VAS 6-point Likert scale (0-5). In total, pain is scored between 0-45 (no pain=0, severe pain=45).
Oswestry Disability Index | Week 0, week 10, week 12
  Disability will be assessed with the Oswestry Disability Index (ODI), which consists of 10 questions that determine functional disability for activities such as sitting, walking, personal care, standing, social life, traveling, and sleeping. Each question has 6 options and the patient is asked to choose the statement that best describes his/her condition. Each question is evaluated between 0-5 points. The question about sexual life may not be answered if it is not appropriate for the person's situation. The higher the score, the higher the level of limitation. The total score percentage varies between 0-100. In scoring, a score of 0-20% indicates minimal disability, 20-40% indicates moderate disability, 40-60% indicates severe disability, and over 60% indicates severe disability. The total score percentage is calculated as follows. "Total Score Percentage= Total Score/(5x Number of Questions Answered) x 100".

SECONDARY OUTCOMES:
Manual Muscle Test | Week 0, week 10, week 12
  Abdominal muscle strength and lumbar extensor muscle strength will be assessed by manual muscle testing as described in the literature.
Pelvic Parameters | Week 0, week 12
  Pelvic parameters (sacral slope angle in degrees, pelvic incidence in degrees, lumbar lordosis in degrees, pelvic tilt in degrees) will be evaluated by the physician on lateral radiographs before treatment and at 3 months. Lateral radiographs will be evaluated in the presence of standard lateral radiographs required for diagnosis and at the 3rd month control, and will not be requested extra from the patients.
Tampa Kinesiophobia Scale | Week 0, week 10, week 12
  Kinesiophobia will be assessed with the 17-item Tampa Kinesiophobia Scale with 4-point Likert scoring. A total score is calculated after reversing items 4, 8, 12 and 16. The person receives a total score between 17-68 and a high score indicates high kinesiophobia.
Global Rating of Change | week 12
  Overall satisfaction and the change perceived by the participants after the training program will be assessed using the Global Rating of Change (GROC). The GROC requires the participant to recall their health status at a time point prior to the intervention and assess their current health status after the intervention, then calculate the difference between the two. The magnitude of this difference is scored by the person on a numeric or visual analog scale. In our study, a numeric scale with descriptive statements at 7 points on it, which is considered reliable in the literature (r = 0.87), will be used.
Use of Orthotics and Home Exercise Diary | On a weekly basis up to 3 months
  The recommended orthotic use and home exercise program will be followed up with daily follow-up. Weekly diary follow-ups will be delivered during the sessions held in the clinic with the therapist and the diary of the new week will be given.

IPD SHARING:
Plan to Share IPD: No